CLINICAL TRIAL: NCT03762018
Title: A Multicentre Randomised Phase III Trial Comparing Atezolizumab Plus Bevacizumab and Standard Chemotherapy Versus Bevacizumab and Standard Chemotherapy as First-line Treatment for Advanced Malignant Pleural Mesothelioma
Brief Title: BEAT-meso: Bevacizumab and Atezolizumab in Malignant Pleural Mesothelioma
Acronym: BEAT-meso
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 13-18; 2018-002180-25 (EudraCT Number); MO40388 (Other: F.Hoffman-La Roche Ltd)
Record Dates: First submitted 2018-11-20; First posted 2018-12-03 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Pleural Mesothelioma Malignant Advanced
Keywords: MPM
MeSH Terms: interventions — Carboplatin; Pemetrexed; Bevacizumab; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bevacizumab plus chemotherapy (Active Comparator): Bevacizumab 15mg/kg intravenously on day 1 every 3 weeks plus 4-6 cycles of carboplatin AUC 5 plus pemetrexed 500mg/m^2 intravenously on day 1 every 3 weeks
  Interventions: Drug: Carboplatin; Drug: Pemetrexed; Drug: Bevacizumab
- Atezolizumab plus bevacizumab plus chemotherapy (Experimental): Atezolizumab 1200mg intravenously on day 1 every 3 weeks plus bevacizumab 15mg/kg intravenously on day 1 every 3 weeks plus 4-6 cycles of carboplatin AUC 5 plus pemetrexed 500mg/m^2 intravenously on day 1 every 3 weeks
  Interventions: Drug: Carboplatin; Drug: Pemetrexed; Drug: Bevacizumab; Drug: Atezolizumab

INTERVENTIONS:
Drug: Carboplatin — Carboplatin belongs to the group of medicines known as alkylating agents. Carboplatin interferes with the growth of cancer cells, which eventually are destroyed.
  Other Names: Carboplatin Accord
Drug: Pemetrexed — Pemetrexed is a type of drug known as an anti metabolite. It stops cells making and repairing DNA so they can't grow and multiply.
  Other Names: Alimta
Drug: Bevacizumab — Bevacizumab is an angiogenesis inhibitor. It works by targeting a protein called vascular endothelial growth factor (VEGF) that helps cancers form new blood vessels. By stopping this process, bevacizumab 'suffocates' the blood supply to the cancer, shrinking it and stopping it from growing.
  Other Names: Avastin
Drug: Atezolizumab — Atezolizumab is in a class of medications called monoclonal antibodies. It works by blocking the action of a certain protein in cancer cells. This helps the immune system to fight against the cancer cells, and helps to slow tumor growth.
  Other Names: Tecentriq; RO5541267
  Arms: Atezolizumab plus bevacizumab plus chemotherapy

SUMMARY:
The aim of this clinical trial is to assess the effect of treatment with a monoclonal antibody called atezolizumab in patients diagnosed with a type of lung cancer called malignant pleural mesothelioma. The efficacy (whether the treatment works), safety and tolerability (side effects of treatment) of atezolizumab plus bevacizumab in combination with standard chemotherapy versus bevacizumab in combination with standard chemotherapy will be investigated.

DETAILED DESCRIPTION:
Malignant pleural mesothelioma (MPM) is a rare and aggressive cancer arising from the mesothelial surface of the pleura. In Europe, the incidence is about 20 per million and is almost always caused by asbestos exposure, with a usual lag time of 30 years between exposure and presentation. Patients diagnosed with advanced MPM have limited treatment options, representing a strict unmet need. Despite decades of clinical research, cytotoxic chemotherapy remains one of the few therapeutic options that has been proven to improve survival in advanced MPM in a randomised controlled trial.

The combination of cisplatin and pemetrexed has become standard first-line therapy worldwide for patients who are not suitable for aggressive surgery or in whom chemotherapy is recommended as part of a multimodality regimen. Carboplatin is often substituted for cisplatin, due to simpler and shorter administration and assumption of a more favourable toxicity profile based on experience in other diseases. Patients with MPM have limited treatment options, representing a strict unmet need.

An antibody is a common type of protein usually made in the body in response to a foreign substance. Antibodies attack foreign substances and protect against infection. The two monoclonal antibodies (atezolizumab and bevacizumab) used in this trial are laboratory-produced antibodies. Atezolizumab is engineered to attach to immune cells to stimulate their activity against cancer cells.

Atezolizumab and bevacizumab are both approved by the European Medicines Agency for the treatment of lung and other cancers. The addition of atezolizumab to bevacizumab plus standard chemotherapy for the treatment of MPM is being investigated in this trial.

All participants will receive 4-6 cycles of standard chemotherapy consisting of carboplatin AUC 5 (area under the plasma concentration versus time curve) plus pemetrexed 500mg/m^2 given intravenously, on day 1 of every 3 week cycle for about 12 to 18 weeks.

Participants will be randomly assigned to one of two treatment groups:

Treatment 1

* Bevacizumab 15 mg/kg intravenously on day 1 of every 3-week cycle, plus
* 4-6 cycles of chemotherapy

OR

Treatment 2

* Atezolizumab 1200 mg fixed dose intravenously on day 1 of every 3-week cycle, plus
* Bevacizumab 15 mg/kg, intravenously on day 1 of every 3-week cycle, plus
* 4-6 cycles of chemotherapy

Participants will continue to receive treatment until disease progression, or until treatment is stopped at the request of the participant or treating doctor, or the participant withdraws consent.

A total of 400 participants from approximately 45 centres in Europe are expected to be included in this trial which will take approximately 6 years to be completed after the first participant is enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced malignant pleural mesothelioma (all histological subtypes are eligible)
* Not amenable for radical surgery based on local standards
* Evaluable disease or measurable disease as assessed according to the modified response evaluation criteria for solid tumours for mesothelioma (mRECIST) v1.1
* Availability of tumour tissue for translational research
* Age >18 years
* Performance Status 0-1
* Life expectancy >3 months
* Adequate haematological, renal and liver function
* Completed baseline quality of life (QoL) questionnaire
* Women of childbearing potential and sexually active men must agree to use highly effective contraception
* Able to understand and give written informed consent and comply with trial procedures

Exclusion Criteria:

* Prior treatment for malignant pleural mesothelioma. Prior radiotherapy for symptom control is allowed, but the irradiated lesion cannot be used as target lesion. If the patient has another target lesion, the patient is eligible.
* Treatment with systemic immune-stimulatory agents within 4 weeks or five half-lives of the drug prior to randomisation and during protocol treatment.
* Treatment with systemic immunosuppressive medications within 2 weeks prior to randomisation and during protocol treatment.
* Previous allogeneic tissue/solid organ transplant
* Live vaccines within 4 weeks prior to first dose of protocol treatment
* Inadequately controlled hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Significant vascular disease within 6 months prior to randomisation
* History of haemoptysis
* Evidence of bleeding diathesis or coagulopathy
* Active autoimmune disease that has required systemic treatment in past 2 years
* History of active diverticulitis
* Previous treatment with atezolizumab and/or bevacizumab or parallel participation in other interventional clinical trial with atezolizumab and/or bevacizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of randomisation until death from any cause, assessed up to 58 months
  Overall survival is defined as the time from the date of randomisation until death from any cause. Data for patients who are not reported as having died at the date of analysis will be censored at the date when they were last known to be alive. Data for patients without post-baseline information will be censored at the date of randomization (plus 1 day).

SECONDARY OUTCOMES:
Progression-free Survival (PFS) according to the mRECIST v1.1 | From date of randomisation until documented progression or death, if progression is not documented, assessed up to 58 months
  PFS is defined as the time from the date of randomisation until documented progression (according to the mRECIST v1.1) or death, if progression is not documented. Censoring (for participants without a PFS/death event) will occur at the date of last tumour assessment. Patients without a post-baseline tumour assessment will be censored at the date of randomization (plus 1 day).
Objective Response Rate (ORR) | From start of protocol treatment acorss all time-points until end of protocol treatment or, as an alternative approach, until the end of follow-up, assessed up to 58 months
  Defined as the percentage of patients that achieve a best overall response [complete response (CR) or partial response (PR)] evaluated according to the mRECIST v1.1 across all post-randomization time-points until the end of protocol treatment or, as an alternative approach, until the end of follow-up. Confirmation of response will not be required.
Disease Control (DC) at 24 weeks | 24 weeks after protocol treatment start
  Defined as complete or partial response, or disease stabilisation at 24 weeks.
Time to Treatment Failure (TTF) | From randomisation until discontinuation of protocol treatment for any reason, assessed up to 58 months
  Defined as the time from the date of randomisation to discontinuation of protocol treatment for any reason (including progression of disease, death, discontinuation of at least one of the drugs consisting the treatment combination due to any reason, such as toxicity or refusal). Censoring will occur at the last follow-up date.
Duration of Response (DoR) | From date of first documentation of objective response until date of first documented progression/ relapse or death, assessed up to 58 months
  Defined as the interval from the date of first documentation of objective response (complete response or partial response, according to the mRECIST v1.1) to the date of first documented progression/ relapse or death.
Number of participants with treatment related adverse events according to Common Toxicity Criteria for Adverse Events (CTCAE) v5.0 | Assessed from the date of informed consent until 90 days after protocol treatment discontinuation. Analysed at 58 months after randomisation of the first patient
  Assessed through analysis of the worst grade of toxicity/adverse events and will include all participants who received at least one dose of protocol treatment. Adverse events leading to dose interruption, withdrawal of protocol treatment and deaths, laboratory parameters and abnormalities and vital signs over the whole treatment period will be assessed and graded according to CTCAE v5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Enriqueta Felip, MD-PhD, Study Chair — Vall d'Hebron University Hospital; Sanjay Popat, PhD, MBBS, Study Chair — Royal Marsden NHS Foundation Trust
Locations (42):
- Belgium (2):
  - University Hospital Leuven, Leuven
  - CHU Liege, Liège
- France (8):
  - Unicancer - Institut Bergonie, Bordeaux
  - Caen- CHU, Caen
  - Le Mans - CHG, Le Mans
  - Lyon - Centre Léon Bérard, Lyon
  - Hospital Nord, Marseille
  - Curie Cancer Center Paris, Paris
  - Toulouse - CHU, Toulouse
  - Tours - CHU, Tours
- Italy (6):
  - SS Antonio e Biagio e Cesare Arrigo Hospital, Alessandria
  - IRCCS Instituto Tumori Giovanni Paolo II, Bari
  - Fondazione IRCCS Istituto Nazionale die Tumori, Milan
  - Instituto Europeo di Oncologia (IEO), Milan
  - AULSS2 Marca Trevigiana Treviso, Treviso
  - University Hospital of Turin, Turin
- Spain (7):
  - Alicante University Hospital ISABIAL, Alicante
  - ICO Hospitalet, Barcelona
  - Vall Hebron University Hospital/Vall Hebron Institue Oncology, Barcelona
  - Puerta de Hierro Hospital, Majadahonda
  - Hospital Parc Tauli Sabadell, Sabadell
  - Virgen del Rocio, Seville
  - Complexo Hospitalario Universitario de Vigo, Vigo
- Switzerland (9):
  - Kantonsspital Aarau, Aarau
  - Istituto Oncologica della Svizzera Italiana, Bellinzona
  - Ferdinando Cerciello, Bern
  - Kantonsspital Graubünden, Chur
  - CHUV, Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - UniversitätSpital Zürich, Zurich
- United Kingdom (10):
  - Addenbrooke's Hospital, Cambridge
  - Clatterbridge Cancer Centre, Liverpool
  - Guy's and St Thomas' Hospital, London
  - Royal Marsden Hospital (Fulham Road), London
  - Royal Marsden Hospital (Sutton), London
  - Kent Oncology Centre, Maidstone
  - Wythenshawe Hospital, Manchester
  - Plymouth Hospitals NHS Trust, Plymouth
  - Weston Park Hospital, Sheffield
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vogelzang NJ, Rusthoven JJ, Symanowski J, Denham C, Kaukel E, Ruffie P, Gatzemeier U, Boyer M, Emri S, Manegold C, Niyikiza C, Paoletti P. Phase III study of pemetrexed in combination with cisplatin versus cisplatin alone in patients with malignant pleural mesothelioma. J Clin Oncol. 2003 Jul 15;21(14):2636-44. doi: 10.1200/JCO.2003.11.136. PMID 12860938
- [Background] Zalcman G, Mazieres J, Margery J, Greillier L, Audigier-Valette C, Moro-Sibilot D, Molinier O, Corre R, Monnet I, Gounant V, Riviere F, Janicot H, Gervais R, Locher C, Milleron B, Tran Q, Lebitasy MP, Morin F, Creveuil C, Parienti JJ, Scherpereel A; French Cooperative Thoracic Intergroup (IFCT). Bevacizumab for newly diagnosed pleural mesothelioma in the Mesothelioma Avastin Cisplatin Pemetrexed Study (MAPS): a randomised, controlled, open-label, phase 3 trial. Lancet. 2016 Apr 2;387(10026):1405-1414. doi: 10.1016/S0140-6736(15)01238-6. Epub 2015 Dec 21. PMID 26719230
- [Background] Ceresoli GL, Zucali PA, Mencoboni M, Botta M, Grossi F, Cortinovis D, Zilembo N, Ripa C, Tiseo M, Favaretto AG, Soto-Parra H, De Vincenzo F, Bruzzone A, Lorenzi E, Gianoncelli L, Ercoli B, Giordano L, Santoro A. Phase II study of pemetrexed and carboplatin plus bevacizumab as first-line therapy in malignant pleural mesothelioma. Br J Cancer. 2013 Aug 6;109(3):552-8. doi: 10.1038/bjc.2013.368. Epub 2013 Jul 16. PMID 23860535
- [Background] Melero I, Berman DM, Aznar MA, Korman AJ, Perez Gracia JL, Haanen J. Evolving synergistic combinations of targeted immunotherapies to combat cancer. Nat Rev Cancer. 2015 Aug;15(8):457-72. doi: 10.1038/nrc3973. PMID 26205340
- [Background] Soto-Ortiz L, Finley SD. A cancer treatment based on synergy between anti-angiogenic and immune cell therapies. J Theor Biol. 2016 Apr 7;394:197-211. doi: 10.1016/j.jtbi.2016.01.026. Epub 2016 Jan 27. PMID 26826488
- [Background] Wallin JJ, Bendell JC, Funke R, Sznol M, Korski K, Jones S, Hernandez G, Mier J, He X, Hodi FS, Denker M, Leveque V, Canamero M, Babitski G, Koeppen H, Ziai J, Sharma N, Gaire F, Chen DS, Waterkamp D, Hegde PS, McDermott DF. Atezolizumab in combination with bevacizumab enhances antigen-specific T-cell migration in metastatic renal cell carcinoma. Nat Commun. 2016 Aug 30;7:12624. doi: 10.1038/ncomms12624. PMID 27571927
- [Background] Tsiouris A, Walesby RK. Malignant pleural mesothelioma: current concepts in treatment. Nat Clin Pract Oncol. 2007 Jun;4(6):344-52. doi: 10.1038/ncponc0839. PMID 17534390
- [Background] Fennell DA, Gaudino G, O'Byrne KJ, Mutti L, van Meerbeeck J. Advances in the systemic therapy of malignant pleural mesothelioma. Nat Clin Pract Oncol. 2008 Mar;5(3):136-47. doi: 10.1038/ncponc1039. PMID 18227828
- [Background] Nowak AK. Chemotherapy for malignant pleural mesothelioma: a review of current management and a look to the future. Ann Cardiothorac Surg. 2012 Nov;1(4):508-15. doi: 10.3978/j.issn.2225-319X.2012.10.05. No abstract available. PMID 23977545
- [Background] Armato SG 3rd, Nowak AK. Revised Modified Response Evaluation Criteria in Solid Tumors for Assessment of Response in Malignant Pleural Mesothelioma (Version 1.1). J Thorac Oncol. 2018 Jul;13(7):1012-1021. doi: 10.1016/j.jtho.2018.04.034. Epub 2018 May 9. PMID 29753121
- [Derived] Uprety D. CheckMate 743: A Glimmer of Hope for Malignant Pleural Mesothelioma. Clin Lung Cancer. 2021 Mar;22(2):71-73. doi: 10.1016/j.cllc.2020.11.009. Epub 2020 Dec 2. No abstract available. PMID 33358660